CLINICAL TRIAL: NCT02542839
Title: Combined Therapy With rTMS and Botulinum Toxin in Primary Cervical Dystonia
Brief Title: rTMS and Botulinum Toxin in Primary Cervical Dystonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: American Brain Foundation (Other); Neuronetics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB201500341
Record Dates: First submitted 2015-06-23; First posted 2015-09-07 (Estimated); Results first posted 2023-09-15 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-08

CONDITIONS: Primary Cervical Dystonia; Dystonia
Keywords: Botulinum Toxin; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Cervical Dystonia, Primary; Dystonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Real rTMS Stimulation (Experimental): Repetitive TMS will be delivered over each cerebellar hemisphere, using a NeuroStar TMS therapy system. The coil will be positioned 3 cm lateral to the inion on the line joining the inion and the external auditory meatus. The coil position will be marked on the skin. 900 pulses will be delivered consecutively to each side with a frequency of 1 Hz and at an intensity of 90% of the resting motor threshold (RMT) for a total duration of 15 min for each cerebellar hemisphere. The RMT will be defined as the lowest stimulation intensity required to evoke a 50 μV potential in a target muscle. Constant coil position will be continuously monitored during the experiment. A similar protocol will be observed for the contralateral cerebellum. In addition, this group will have the following performed: Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) test, Cerebellar-brain Inhibition (CBI) measurement, and Craniocervical Dystonia Questionnaire (CDQ-24) questionnaire to fill out.
  Interventions: Device: NeuroStar TMS therapy; Other: Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS); Other: Craniocervical Dystonia Questionnaire (CDQ-24); Other: Cerebellar-brain Inhibition (CBI); Procedure: Botulinum toxin injections
- Sham rTMS Stimulation (Sham Comparator): Patients will undergo the same procedure for identifying stimulus location used in patients receiving real rTMS. Simulated rTMS will be administered using sham NeuroStar TMS therapy system coil which produces discharge noise and vibration without stimulating the cerebral cortex. This technique has been suggested to provide more effective blinding compared to other methods use in previous controlled studies. In addition, this group will have the following performed: Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) test, Cerebellar-brain Inhibition (CBI) measurement, and Craniocervical Dystonia Questionnaire (CDQ-24) questionnaire to fill out.
  Interventions: Device: Sham NeuroStar TMS therapy; Other: Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS); Other: Craniocervical Dystonia Questionnaire (CDQ-24); Other: Cerebellar-brain Inhibition (CBI); Procedure: Botulinum toxin injections

INTERVENTIONS:
Device: NeuroStar TMS therapy — Application of repetitious transcranial magnetic stimulation (TMS) pulses using NeuroStar device to a specific brain target at predefined stimulation parameters.
  Arms: Real rTMS Stimulation
Device: Sham NeuroStar TMS therapy — Same procedure as real rTMS without stimulating the cerebral cortex.
  Arms: Sham rTMS Stimulation
Other: Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) — All participants will receive a clinical assessment of dystonia severity by using the TWSTRS test.
Other: Craniocervical Dystonia Questionnaire (CDQ-24) — All participants will fill out the Craniocervical Dystonia Questionnaire (CDQ-24) quality of life questionnaire.
Other: Cerebellar-brain Inhibition (CBI) — All participants will have a measure of the cerebellar-brain inhibition(CBI) which will be conducted by using a TMS device determining the ability of the coil to activate the cerebellum.
Procedure: Botulinum toxin injections — All participants will receive Botulinum toxin(BoNT) injections as part of their standard of care

SUMMARY:
Primary cervical dystonia (PCD) is the most common form of focal dystonia. PCD is frequently reported as a source of disability, decreased quality of life, and social stigma. Botulinum toxin (BoNT) is the gold standard treatment for PCD. The average duration of benefits from BoNT injections was about 9.5 weeks and BoNT treatment is known to provide only pure symptomatic benefits and does not seem to modify the disease pathophysiology.

The investigator plans to use repetitive transcranial magnetic stimulation (rTMS) therapy as an adjunctive therapy in combination with BoNT injections as a novel approach to treat PCD. The primary goal of this study is to compare standard treatment with BoNT versus BoNT combined with a two week course of rTMS.

DETAILED DESCRIPTION:
rTMS refers to the application of transcranial magnetic stimulation (TMS) pulses to a specific target at predefined stimulation parameters. Repeated sessions of rTMS therapy have been demonstrated to induce cumulative persistent benefits that can last weeks after the conclusion of the rTMS sessions

The central hypothesis of this study is that rTMS therapy in PCD can potentiate the effects of BoNT injections. With the current standard treatment, the peak-dose benefits seen with BoNT are seen at about 4-6 weeks after the administration of injections. The investigator will introduce a 1 week course of rTMS around 2-8 weeks before or after BoNT or T1). The investigator will examine the effects of combined therapy at 10 weeks after BoNT and 12 weeks after BoNT injections follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCD in accordance with the Consensus Statement of the Movement Disorder Society
* Subjects who report Botulinum Toxin benefits lasting 10 weeks or less only (suboptimal benefits with standard care)

Exclusion Criteria:

* Pregnancy
* Active seizure disorder
* Presence of a metallic body such as pacemaker, implants, metal rods and hearing aid.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Wagle-Shukla, M.D., Principal Investigator — UF Center for Movement Disorders and Neurorestoration
Locations (2):
- United States (2):
  - UF Center for Movement Disorders & Neurorestoration, Gainesville, Florida
  - UF Brain Institute, Gainesville, Florida

REFERENCES:
- [Background] Tarsy D, Simon DK. Dystonia. N Engl J Med. 2006 Aug 24;355(8):818-29. doi: 10.1056/NEJMra055549. No abstract available. PMID 16928997
- [Background] Phukan J, Albanese A, Gasser T, Warner T. Primary dystonia and dystonia-plus syndromes: clinical characteristics, diagnosis, and pathogenesis. Lancet Neurol. 2011 Dec;10(12):1074-85. doi: 10.1016/S1474-4422(11)70232-0. Epub 2011 Oct 24. PMID 22030388
- [Background] Jankovic J. Treatment of dystonia. Lancet Neurol. 2006 Oct;5(10):864-72. doi: 10.1016/S1474-4422(06)70574-9. PMID 16987733
- [Background] Dressler D, Tacik P, Saberi FA. Botulinum toxin therapy of cervical dystonia: duration of therapeutic effects. J Neural Transm (Vienna). 2015 Feb;122(2):297-300. doi: 10.1007/s00702-014-1253-8. Epub 2014 Jul 23. PMID 25052566
- [Background] Thenganatt MA, Jankovic J. Treatment of dystonia. Neurotherapeutics. 2014 Jan;11(1):139-52. doi: 10.1007/s13311-013-0231-4. PMID 24142590
- [Background] Hallett M. Transcranial magnetic stimulation: a primer. Neuron. 2007 Jul 19;55(2):187-99. doi: 10.1016/j.neuron.2007.06.026. PMID 17640522
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Wagle Shukla A, Vaillancourt DE. Treatment and physiology in Parkinson's disease and dystonia: using transcranial magnetic stimulation to uncover the mechanisms of action. Curr Neurol Neurosci Rep. 2014 Jun;14(6):449. doi: 10.1007/s11910-014-0449-5. PMID 24771105
- [Background] Rossi S, Ferro M, Cincotta M, Ulivelli M, Bartalini S, Miniussi C, Giovannelli F, Passero S. A real electro-magnetic placebo (REMP) device for sham transcranial magnetic stimulation (TMS). Clin Neurophysiol. 2007 Mar;118(3):709-16. doi: 10.1016/j.clinph.2006.11.005. Epub 2006 Dec 22. PMID 17188568

RESULTS

PARTICIPANT FLOW:
Groups:
- Real rTMS Stimulation: Repetitive TMS will be delivered over each cerebellar hemisphere, using a NeuroStar TMS therapy system. The coil will be positioned 3 cm lateral to the inion on the line joining the inion and the external auditory meatus. The coil position will be marked on the skin. 900 pulses will be delivered consecutively to each side with a frequency of 1 Hz and at an intensity of 90% of the resting motor threshold (RMT) for a total duration of 15 min for each cerebellar hemisphere. The RMT will be defined as the lowest stimulation intensity required to evoke a 50 μV potential in a target muscle. Constant coil position will be continuously monitored during the experiment. A similar protocol will be observed for the contralateral cerebellum.
  NeuroStar TMS therapy: Application of repetitious transcranial magnetic stimulation (TMS) pulses using NeuroStar device to a specific brain target at predefined stimulation parameters.
  Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS): All participants will receive a clinical assessment of dystonia severity by using the TWSTRS test.
  Craniocervical Dystonia Questionnaire (CDQ-24): All participants will fill out the Craniocervical Dystonia Questionnaire (CDQ-24) quality of life questionnaire.
  Cerebellar-brain Inhibition (CBI): All participants will have a measure of the cerebellar-brain inhibition(CBI) which will be conducted by using a TMS device determining the ability of the coil to activate the cerebellum.
Period: Overall Study
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Real rTMS Stimulation: Repetitive TMS will be delivered over each cerebellar hemisphere, using a NeuroStar TMS therapy system. The coil will be positioned 3 cm lateral to the inion on the line joining the inion and the external auditory meatus. The coil position will be marked on the skin. 900 pulses will be delivered consecutively to each side with a frequency of 1 Hz and at an intensity of 90% of the resting motor threshold (RMT) for a total duration of 15 min for each cerebellar hemisphere.
  NeuroStar TMS therapy: Application of repetitious transcranial magnetic stimulation (TMS) pulses using NeuroStar device to a specific brain target at predefined stimulation parameters.
  Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS): All participants will receive a clinical assessment of dystonia severity by using the TWSTRS test.
  Craniocervical Dystonia Questionnaire (CDQ-24): All participants will fill out the Craniocervical Dystonia Questionnaire (CDQ-24) quality of life questionnaire.
  Cerebellar-brain Inhibition (CBI): All participants will have a measure of the cerebellar-brain inhibition(CBI) which will be conducted by using a TMS device determining the ability of the coil to activate the cerebellum.
  Botulinum toxin injections: All participants will receive Botulinum toxin(BoNT) injections as part of their standard of care
- Total: Total of all reporting groups
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (6) | 59 (6) | 60 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Dystonia Severity as Assessed by the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS)
Description: A clinical assessment of dystonia severity will be conducted at each study visit using the TWSTRS. The TWSTRS is a widely accepted composite rating scale for PCD with subscales for clinical severity, functional disability, and associated pain. The total score reported here can range 0-85, where a higher scores represent greater dystonia severity.
Time Frame: absolute value at 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
Number analyzed (Participants) | 5 | 4
scores on a scale | 13 (6) | 17 (8)

2. Secondary Outcome: TMS Measure Referred to as Cerebellar Inhibition (CBI)
Description: A measure of the cerebellar-brain inhibition(CBI) will be conducted using a TMS device determining the ability of the coil to activate the cerebellum. CBI is calculated by taking the mean of amplitudes of motor-evoked potentials (mV) in response to conditioned stimulation and dividing it by the mean of amplitudes of motor-evoked potentials (mV) in response to unconditioned stimulation (i.e., the control condition). Thus it is a measure of the degree of inhibition due to a conditioning stimulus, where <1 indicates inhibition, =1 indicates no inhibition, and >1 indicates not inhibition but excitation. As a ratio of amplitudes, it does not have units.
Time Frame: absolute value at 12 weeks
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Real rTMS Stimulation: Repetitive TMS will be delivered over each cerebellar hemisphere, using a NeuroStar TMS therapy system. The coil will be positioned 3 cm lateral to the inion on the line joining the inion and the external auditory meatus. The coil position will be marked on the skin. 900 pulses will be delivered consecutively to each side with a frequency of 1 Hz and at an intensity of 90% of the resting motor threshold (RMT) for a total duration of 15 min for each cerebellar hemisphere. The RMT will be defined as the lowest stimulation intensity required to evoke a 50 μV potential in a target muscle.
  NeuroStar TMS therapy: Application of repetitious transcranial magnetic stimulation (TMS) pulses using NeuroStar device to a specific brain target at predefined stimulation parameters.
  Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS): All participants will receive a clinical assessment of dystonia severity by using the TWSTRS test.
  Craniocervical Dystonia Questionnaire (CDQ-24): All participants will fill out the Craniocervical Dystonia Questionnaire (CDQ-24) quality of life questionnaire.
  Cerebellar-brain Inhibition (CBI): All participants will have a measure of the cerebellar-brain inhibition(CBI) which will be conducted by using a TMS device determining the ability of the coil to activate the cerebellum.
  Botulinum toxin injections: All participants will receive Botulinum toxin(BoNT) injections as part of their standard of care
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
Number analyzed (Participants) | 5 | 4
ratio | 0.7 (0.2) | 0.9 (0.3)

3. Secondary Outcome: Craniocervical Dystonia Questionnaire
Description: The Craniocervical Dystonia Questionnaire (CDQ-24) is a patient-rated health related quality of life (HR-QoL) measure for craniocervical dystonia. It is composed of 24 items, forming 5 subscales: stigma, emotional well-being, pain, activities of daily living, and social/ family life. Items are rated on a 5-point scale. Each item consists of five statements representing increasing severity of impairment, scored from 0 to 4. Subjects will be instructed to indicate how they have felt during the past two weeks because of dystonia by selecting one of the five statements for each item. The total score reported here can range from 0-96, with a higher score indicating a greater impact of dystonia on quality of life.
Time Frame: absolute value at 12 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Real rTMS Stimulation: Repetitive TMS will be delivered over each cerebellar hemisphere, using a NeuroStar TMS therapy system. The coil will be positioned 3 cm lateral to the inion on the line joining the inion and the external auditory meatus. The coil position will be marked on the skin. 900 pulses will be delivered consecutively to each side with a frequency of 1 Hz and at an intensity of 90% of the resting motor threshold (RMT) for a total duration of 15 min for each cerebellar hemisphere. The RMT will be defined as the lowest stimulation intensity required to evoke a 50 μV potential in a target muscle.
  Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS): All participants will receive a clinical assessment of dystonia severity by using the TWSTRS test.
  Craniocervical Dystonia Questionnaire (CDQ-24): All participants will fill out the Craniocervical Dystonia Questionnaire (CDQ-24) quality of life questionnaire.
  Cerebellar-brain Inhibition (CBI): All participants will have a measure of the cerebellar-brain inhibition(CBI) which will be conducted by using a TMS device determining the ability of the coil to activate the cerebellum.
  Botulinum toxin injections: All participants will receive Botulinum toxin(BoNT) injections as part of their standard of care
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
Number analyzed (Participants) | 5 | 4
score on a scale | 16 (4) | 18 (6)

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Sham rTMS Stimulation: Patients will undergo the same procedure for identifying stimulus location used in patients receiving real rTMS. Simulated rTMS will be administered using sham NeuroStar TMS therapy system coil which produces discharge noise and vibration without stimulating the cerebral cortex.
  Sham NeuroStar TMS therapy: Same procedure as real rTMS without stimulating the cerebral cortex.
  Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS): All participants will receive a clinical assessment of dystonia severity by using the TWSTRS test.
  Craniocervical Dystonia Questionnaire (CDQ-24): All participants will fill out the Craniocervical Dystonia Questionnaire (CDQ-24) quality of life questionnaire.
  Cerebellar-brain Inhibition (CBI): All participants will have a measure of the cerebellar-brain inhibition(CBI) which will be conducted by using a TMS device determining the ability of the coil to activate the cerebellum.
  Botulinum toxin injections: All participants will receive Botulinum toxin(BoNT) injections as part of their standard of care
Arm/Group | Real rTMS Stimulation | Sham rTMS Stimulation
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 2/5 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real rTMS Stimulation (N=5) | Sham rTMS Stimulation (N=4)
headaches (Nervous system disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT02542839/Prot_SAP_000.pdf